CLINICAL TRIAL: NCT06884839
Title: Tumor Deposits in Colorectal Cancer and Its Prognostic Value in Survival and Metastasis
Status: Recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Salah, Lecturer of General Surgery, Faculty of Medicine, Minia University, Minia, Egypt., Minia University
Other Study IDs: 1267/09/2024
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Tumor Deposits; Colorectal Cancer; Prognosis; Survival; Metastasis
MeSH Terms: conditions — Extranodal Extension; Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Therapeutic resection group: Patients with colorectal cancer underwent therapeutic resection with pathologically positive tumor deposits (TDs) to determine distant metastasis occurrence and the effect of TDs on survival.
  Interventions: Procedure: Therapeutic resection

INTERVENTIONS:
Procedure: Therapeutic resection — Patients with colorectal cancer underwent therapeutic resection with pathologically positive tumor deposits (TDs) to determine distant metastasis occurrence and the effect of TDs on survival.

SUMMARY:
This study aims to evaluate the tumor deposits in colorectal cancer and its prognostic value in survival and metastasis

DETAILED DESCRIPTION:
Tumor deposits (TDs) are defined as isolated tumor foci found in the pericolonic or perirectal fat or the adjacent mesentery (mesocolonic fat) away from the invasive margin of the tumor without evidence of residual lymphatic tissue. TDs are significantly correlated with poor prognosis after colorectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old.
* Both sexes.
* All Colorectal cancer patients From Stage I to III Colorectal cancer with pathologically positive Tumor deposits.

Exclusion Criteria:

* Patient took neoadjuvant therapy.
* No information available on tumor deposits.
* Colorectal cancer is not the only primary cancer.
* Patients with incomplete information about follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective and retrospective study will be conducted on 30 patients with colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Patients' overall survival | 2 years postoperatively
  Patients' overall survival (OS) is defined as from colorectal cancer (CRC) diagnosis to death.

SECONDARY OUTCOMES:
Distant metastasis | 2 years postoperatively
  Distant metastasis is defined as the presence of liver, lung, bone, or brain metastases during or after colorectal cancer (CRC) diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.